CLINICAL TRIAL: NCT04858204
Title: Real Life Second-Line Nivolumab in Advanced Non-Small Cell Lung Cancer: a French Observational Multicenter Study of 259 Patients (ABCT-IMMUNOBZH)
Brief Title: Real Life Second-Line Nivolumab in Advanced Non-Small Cell Lung Cancer
Acronym: IMMUNOBZH
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMMUNOBZH (29BRC17.0032)
Record Dates: First submitted 2018-09-13; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2017-04

CONDITIONS: NSCLC
Keywords: Real-life; nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data regarding nivolumab as second line treatment in advanced non-small cell lung cancer (NSCLC) are based on selected populations and might not reflect daily practice. Investigators aimed at assessing efficacy and safety of nivolumab in a real-life setting and determining a subtype of NSCLC patients that are more likely to benefit from immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* advanced NSCLC (stage IIIB-IV)
* failure of at least one line of chemotherapy.
* age ≥18 years,
* initiation of nivolumab between 01/09/2015 and 30/09/2016.

Exclusion Criteria:

* nivolumab initiation after October 2016
* prior involvement in an immunotherapy trial
* refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced stage non-small cell lung cancer patients
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Nivolumab Objective response rate | through study completion, an average of 1 year
  Objective response rate evaluated by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHRU de Brest, Brest
  - CH DINAN, Dinan
  - Centre Hospitalier de Bretagne Sud, Lorient
  - CHU de Rennes, Rennes
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Centre hospitalier de Saint Malo, St-Malo
  - CH de VANNES, Vannes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Malhotra J, Jabbour SK, Aisner J. Current state of immunotherapy for non-small cell lung cancer. Transl Lung Cancer Res. 2017 Apr;6(2):196-211. 2. Kazandjian D, Suzman DL, Blumenthal G, Mushti S, He K, Libeg M et al. FDA Approval Summary: Nivolumab for the Treatment of Metastatic Non-Small Cell Lung Cancer With Progression On or After Platinum-Based Chemotherapy. The Oncologist. 2016 May;21(5):634-42. 3. Brahmer J, Reckamp KL, Baas P, Crinò L, Eberhardt WE, Poddubskaya E et al. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. 4. Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE et al. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. 5. Herbst RS, Baas P, Kim D-W, Felip E, Pérez-Gracia JL, Han JY et al. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. The Lancet. 2016 Apr;387(10027):1540-50. 6. Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J et al. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet Lond Engl. 2017 21;389(10066):255-65. 7. Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer Oxf Engl 1990. 2009 Jan;45(2):228-47. 8. Common Terminology Criteria for Adverse Events (CTCAE) - CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf